CLINICAL TRIAL: NCT04236765
Title: Tuberculosis Infection in Children Visiting Friends and Relatives in Countries With High Incidence of Tuberculosis: a Study Protocol
Brief Title: Tuberculosis In Children Visiting Friends and Relatives
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Mutua de Terrassa (Other)
Collaborators: Public Health Agency of Barcelona (Other); Hospital Vall d'Hebron (Other); Hospital Sant Joan de Deu (Other); Institut Català de la Salut (Other); Hospital Universitari Sant Joan de Reus (Other); Hospital de Tortosa Verge de la Cinta (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: P16/094
Record Dates: First submitted 2020-01-10; First posted 2020-01-22 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Tuberculosis Infection
Keywords: Tuberculosis; Latent Tuberculosis; Children; Immigrant; Incidence; Travel-Related Infection; Tuberculin Test; Interferon-gamma Release Assay
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis; Travel-Related Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TB infection-screening benefiting group (Experimental): children VFRs under 15 years of age (which are children of immigrants and born or not in Spain) who travel to countries with an elevated incidence of TB will be screened for LTBI after their return.
  Interventions: Other: TB infection-screening benefiting group

INTERVENTIONS:
Other: TB infection-screening benefiting group — The children who participate in the study will be recruited during a programmed visit to a traveler health clinic or a primary care center. During the first visit the parents or legal guardian will be interviewed, a questionnaire will be completed with sociodemographic, epidemiologic and clinical data and a tuberculin skin test (TST) will be performed and read at 48-72 hours. At 8-12 weeks after returning from the travel abroad the child will have a new visit. A new interview will be carried out with the parents or legal guardian and a questionnaire will be completed with epidemiological and clinical data. The child will undergo a new TST and QFT-Plus test.

SUMMARY:
In countries with a low incidence of Tuberculosis (TB), the incidence remains higher among the immigrant population than among the autochthonous population beyond the first years after arrival in the host country. In addition, at a pediatric level, most cases are produced in immigrant children and the children of immigrants. This persistence of a greater incidence in the immigrant population might, in part, be explained by the increase in exposure to Mycobacterium tuberculosis during trips to their country of origin to visit friends and relatives (VFRs). The objectives of the study are to estimate the risk of latent infection by M. tuberculosis (LTBI)/TB in children VFRs and the factors associated with this risk. The investigators will also study the behavior of the diagnostic tests. This project will be carried out in collaboration with 21 primary health care centers and 5 hospitals in Catalonia.

DETAILED DESCRIPTION:
A prospective study will be carried out. The study subjects are children under 15 years of age, which are children of immigrants and born or not in Spain, who travel to VFRs to countries with an elevated incidence of TB (> 40 cases/100,000 inhabitants). A sample size of 492 children was estimated. Children will be recruited during a programmed visit to a traveler health clinic or a primary care center, a questionnaire will be completed with sociodemographic, epidemiologic and clinical data and a tuberculin skin test (TST) will be performed and read at 48-72 hours. At 8-12 weeks after returning from the travel abroad the child will have a new visit in which a questionnaire will be completed with epidemiological and clinical data, an a TST and QFT-Plus test will be performed. The rate of incidence of LTBI will be estimated per individual/month and person/year per country visited and by age group.

ELIGIBILITY:
Inclusion Criteria (all criteria must be met):

* Informed consent must be obtained from the parents of legal guardian.
* Less than 15 years of age.
* One or both of the parents is from a country with an elevated incidence of TB. A country is considered to have an elevated incidence of TB when this incidence is 3-fold higher than the incidence in Catalunya, that is approximately 40/100,000 inhabitants. Countries with official reports describing an incidence less than the value proposed but which have regions with > 40 cases /100,000 inhabitants are also included (Table and figure 1)
* The journey to the country of origin is made by at least one of the parents.
* The duration of the visit to the country of origin is of at least 21 days.

Exclusion Criteria:

* Previous TB or LTBI.
* Tourist visit to hotels and resorts with scarce contact with the autochthonous population.
* Primary or secondary immunodeficiency to treatment with corticosteroids, transplantation, treatment with anti-tumor necrosis factor, chronic renal insufficiency.
* Congenital cardiopathy.
* Cystic fibrosis of the pancreas and other congenital diseases of pulmonary origin.

Ages: 6 Months to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 492 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
change in health status: LTBI diagnosis after having traveled abroad | At 8-12 weeks after returning from the travel abroad
  To be evaluated with Tuberculin test and Interferon-gamma release assay (QuantiFERON-TB Gold Plus (QFT-Plus)). LTBI is defined as having at least one positive infection test (Tuberculin Test and/or QFT-Plus)

SECONDARY OUTCOMES:
Sociodemographic characteristics of the patients | baseline (before traveling abroad)
  sex, date of birth, country of child's birth, country of father's and mother's birth.
  To be evaluated with an ad hoc questionnaire.
Epidemiological data (before travel abroad): | baseline (before travel abroad)
  history of previous study for tuberculosis infection, pre-travel visit date, country of trip, probable travel date.
  To be evaluated with an ad hoc questionnaire.
Epidemiological data (after travel abroad): | At 8-12 weeks after returning from the travel abroad
  travel date, post-travel visit date, return date of the trip, travel time, number of cohabitants at the address visited, travel environment (rural / urban / mixed), smokers in the home visited.
  To be evaluated with an ad hoc questionnaire.
Clinical data: Bacillus Calmette-Guerin (BCG) vaccination | baseline (before travel abroad)
  Bacillus Calmette-Guerin (BCG) vaccination (yes/no type). To be evaluated with an ad hoc questionnaire.
Clinical data: presence of BCG scar | baseline (before travel abroad)
  presence of BCG scar (yes/no type). To be evaluated with an ad hoc questionnaire.
Clinical data: height | baseline (before travel abroad) and follow-up (At 8-12 weeks after returning from the travel abroad )
  height in meters. To be evaluated with an ad hoc questionnaire.
Clinical data: weight | baseline (before travel abroad) and follow-up (At 8-12 weeks after returning from the travel abroad )
  weight in kilograms. To be evaluated with an ad hoc questionnaire. To be evaluated with an ad hoc questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Mutua Terrassa, Terrassa, Barcelona, Spain

REFERENCES:
- [Derived] Soriano-Arandes A, Cayla JA, Goncalves AQ, Orcau A, Noguera-Julian A, Padilla E, Sola-Segura E, Gordillo NR, Espiau M, Garcia-Lerin MG, Rifa-Pujol MA, Jordi Gomez I Prat, Macia-Rieradevall E, Martin-Nalda A, Eril-Rius M, Santos Santiago J, Busquets-Poblet L, Martinez RM, Perez-Porcuna TM. Tuberculosis infection in children visiting friends and relatives in countries with high incidence of tuberculosis: A study protocol. Medicine (Baltimore). 2020 Sep 4;99(36):e22015. doi: 10.1097/MD.0000000000022015. PMID 32899054